CLINICAL TRIAL: NCT01453868
Title: The Effects of Neuromuscular Training on Balance in Patients With Multiple Sclerosis
Brief Title: The Effects of Aerobics Training on Balance in Patients With Multiple Sclerosis
Acronym: NIA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nelson Mandela Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr. Donovan Adendorf, Dr Donovan Adendorf, Nelson Mandela Metropolitan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H11-HEA-HMS-002
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; non impact aerobics
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active non impact aerobics (Active Comparator): This group will be performing a 12 week non impact aerobics program twice a week.
  Interventions: Other: Non Impact Aerobics
- Control group: Passive lecture series (Active Comparator): The control group will also be measured for balance and then attend a 12 week lecture series with no exercise. They will then also be remeasured post lectures series
  Interventions: Other: Passive : lecture series

INTERVENTIONS:
Other: Non Impact Aerobics — a 12 week, twice a week class in non impact aerobics
  Other Names: Dancing, NIA, MS
  Arms: Active non impact aerobics
Other: Passive : lecture series — a 12 week, once a week for one hour lecture series with no exercise. Topics will cover symptom management in Multiple Sclerosis
  Other Names: Lifestyle lectures, symptom management
  Arms: Control group: Passive lecture series

SUMMARY:
Standing Balance, with and without blindfold, will be measured on patients with Multiple Sclerosis using a Biodex Balance Scale.

A Twelve week intervention with one non impact aerobics group and one control group will be performed.

Standing balance will then be retested on all subjects and the results will be statistically compared.

DETAILED DESCRIPTION:
Standing Balance will be tested in 4 phases:

* On a firm surface eyes open
* On a frim surface eyes blindfolded
* On a foam surface eyes open
* On a foam surface eyes blindfolded

The aerobics classes will be conducted by a NIA (Non Impact Aerobics) instructor and will be a combination of tai chi, slow movement dancing, stretching and modified yoga stretches.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were diagnosed by a neurologist with Relapsing Remitting Multiple Sclerosis.
* EDSS scale between 1 and 6.
* Patients that are able to travel to and from a 12 week program location.

Exclusion Criteria:

* Patients that were diagnosed by a neurologist with primary or secondary progressive multiple sclerosis.
* EDSS scale above 6

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Biodex Scale Balance score: Automated | Change: baseline and 12 weeks
  A patient will step up to a Biodex Balance scale and will be instructed to try and maintain balance on the machine until it produces an automated outcome score for balance. This number is directly related to a fall risk score in patients with neurological compromise.

SECONDARY OUTCOMES:
Pre and post intervention questionaire | Change: baseline and 12 weeks
  A fifty question questionaire will be administered pre and post intervention. These questions will focus on mood changes, attitude changes and overall quality of life changes related to adding exercise in their daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Donovan Adendorf, DC, Principal Investigator — Nelson Mandela Metropole University, Department of Health Sciences; Rosa DuRandt, PhD, Study Director — Professor: Human Movement Sciences, NMMU-Port Elizabeth South Africa; Maryna Baard, PhD, Study Chair — Faculty of Helath Sciences-NMMU, Port Elizabeth South Africa
Locations (1):
- HealthZone Chiropractic Clinic, Gaylord, Michigan, United States

REFERENCES:
- See also: Nelson Mandela Metropole University, Port Elizabeth South Africa — http://www.nmmu.ac.za/